CLINICAL TRIAL: NCT01081236
Title: The Role of the Intestinal Barrier Function in Liver Cirrhosis
Brief Title: Intestinal Barrier Function and Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. dr. A. Masclee, Maastricht University Medical Center, Division of Gastroenterology-Hepatology
Other Study IDs: MEC 09-2-125
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-12

CONDITIONS: Liver Cirrhosis
Keywords: liver cirrhosis; intestinal permeability; microbiota; complications
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Compensated liver cirrhosis
- Decompensated liver cirrhosis

SUMMARY:
Patients with liver cirrhosis have an increased risk to develop life-threatening complications such as spontaneous bacterial peritonitis (SBP). Impairment in the intestinal barrier, changes in numbers and composition of the intestinal microbiota and alterations in immune defenses have been suggested to be involved in liver cirrhosis and its complications. Dysfunction in the intestinal barrier for example results in the ongoing passage of toxic substances from the gastrointestinal tract that may damage the liver, leading to oxidative stress, inflammation and eventually liver cirrhosis. In addition, bacterial translocation is considered a key step in the development of spontaneous infections, mainly SBP, in patients with liver cirrhosis.

The investigators hypothesize that patients with decompensated liver cirrhosis have a more impaired intestinal epithelial barrier and altered intestinal microbiota than patients with compensated liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis of any cause
* A score of greater-than or equal to 5 assessed according to the Child-Pugh classification
* Age between 18 and 65 years

Exclusion Criteria:

* Known gastrointestinal diseases (such as inflammatory bowel disease and celiac disease), chronic renal disease (i.e. a glomerular filtration rate of less-than or equal to 60 ml/min per 173 m2 estimated from the Modification of Diet in Renal Disease (MDRD) equation) or Diabetes Mellitus
* Major abdominal surgery interfering with gastrointestinal function (except for uncomplicated appendectomy, cholecystectomy and hysterectomy, other surgery upon judgement of the principle investigator)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be selected from a hospital providing both secondary and tertiary care
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The primary aim is to study differences in small and large intestinal permeability between patients with compensated and decompensated cirrhosis by means of a sugar permeability test | 2 years

SECONDARY OUTCOMES:
To assess tight junction structure and proteins in biopsy specimens of small and large intestine | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: A Masclee, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands